CLINICAL TRIAL: NCT04624659
Title: An Adaptive, Randomized, Placebo-controlled, Double-blind, Multi-center Study of Oral Etavopivat, a Pyruvate Kinase Activator in Patients With Sickle Cell Disease (HIBISCUS)
Brief Title: A Study of Etavopivat in Adults and Adolescents With Sickle Cell Disease (HIBISCUS)
Acronym: HIBISCUS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Forma Therapeutics, Inc. (Industry)
Collaborators: This study is currently undergoing a sponsor transition from Forma to Novo Nordisk. Sponsor field will be updated once the transition is complete. (Unknown)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4202-HEM-301
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Sickle Cell; Anemia; Sickle Cell Anemia; Hemolytic; Hemoglobin; Vaso-occlusive Crisis; Sickle Cell Crisis; Congenital Anemia; Hemolytic Anemia; Hematologic Disease; Hemoglobinopathies; Genetic Disease; Inborn Disease; Sickle Cell Trait; Pyruvate Kinase
MeSH Terms: conditions — Anemia, Sickle Cell; Anemia; Hemolysis; Vaso-Occlusive Crises; Anemia, Hemolytic; Hematologic Diseases; Hemoglobinopathies; Genetic Diseases, Inborn; Sickle Cell Trait

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Double blind etavopivat Low Dose (Experimental): Double blind etavopivat Low Dose
  Interventions: Drug: Etavopivat Tablets Low dose
- Double blind etavopivat High Dose (Experimental): Double blind etavopivat High Dose
  Interventions: Drug: Etavopivat Tablets High dose
- Double blind placebo (Experimental): Double blind placebo
  Interventions: Drug: Placebo Tablets
- Open label etavopivat (Experimental): Open label etavopivat
  Interventions: Drug: Etavopivat Tablets

INTERVENTIONS:
Drug: Etavopivat Tablets Low dose — 200 mg once daily
  Other Names: FT-4202
  Arms: Double blind etavopivat Low Dose
Drug: Etavopivat Tablets High dose — 400 mg once daily
  Other Names: FT-4202
  Arms: Double blind etavopivat High Dose
Drug: Placebo Tablets — Placebo once daily
  Other Names: placebo
  Arms: Double blind placebo
Drug: Etavopivat Tablets — Selected dose once daily
  Other Names: FT-4202
  Arms: Open label etavopivat

SUMMARY:
This clinical trial is a Phase 2/3 study that will evaluate the efficacy and safety of etavopivat and test how well etavopivat works compared to placebo to improve the amount of hemoglobin in the blood and to reduce the number of vaso-occlusive crises (times when the blood vessels become blocked and cause pain).

DETAILED DESCRIPTION:
Etavopivat is designed to activate PKR and thereby modulate RBC metabolism by impacting two critical pathways in RBCs. The etavopivat clinical development program will investigate whether decreasing 2,3-DPG may help oxygen bind to hemoglobin (i.e. increasing oxygen affinity), and thereby increase ATP and impact RBC function. This study is a randomized, placebo-controlled, double-blind, multicenter Phase 2/3 study of patients age 12 to 65 years (inclusive), with sickle cell disease. There is one planned interim analyses in this study design. Initially, patients will be randomized at 1:1:1 to one of two dose levels of etavopivat or placebo. At the first interim analysis, one of the two etavopivat dose levels will be selected for the Phase 3 portion of the study, in which patients will be randomized at 1:1 to the selected etavopivat dose or placebo. Efficacy on hemoglobin will be evaluated at conclusion of the double-blind treatment period. Following completion of 52 weeks of double-blind treatment, patients may enter a 112-week etavopivat open-label extension period.

ELIGIBILITY:
Key Inclusion Criteria:

* Provision of consent
* Patient has a confirmed diagnosis of sickle cell disease
* At least 2 episodes of vaso-occlusive crises in the past 12 months
* Hemoglobin ≥ 5.5 and ≤ 10.5 g/dL (≥ 55 and ≤ 105 g/L) during screening
* Patients taking hydroxyurea, must demonstrate a stable dose for at least 90 days prior to start of study treatment
* Patients on crizanlizumab or L-glutamine treatment at the time of consent must be on a stable dose for ≥ 12 months and must be ≥ 80% compliant with the planned regimen at the time of consent and meet the VOC eligibility criteria
* Female patients of childbearing potential must use highly effective methods of contraception, male patients are willing to use barrier methods of contraception

Key Exclusion Criteria:

* More than 15 vaso-occlusive crises within the past 12 months
* Female who is breastfeeding or pregnant
* Hepatic dysfunction characterized by:

  * Alanine aminotransferase (ALT) > 4.0 × upper limit of normal (ULN)
  * Direct bilirubin > 3.0 × ULN
* Known HIV positivity
* Active hepatitis B or hepatitis C infection
* Severe renal dysfunction or on chronic dialysis
* History of unstable or deteriorating cardiac or pulmonary disease within 6 months prior to consent including but not limited to the following:

  * Unstable angina pectoris or myocardial infarction or elective coronary intervention
  * Congestive heart failure requiring hospitalization
  * Uncontrolled clinically significant arrhythmias
  * Symptomatic pulmonary hypertension
* History of overt clinical stroke within previous 2 years or any history of an intracranial hemorrhage
* History of deep venous thrombosis requiring systemic anti-coagulation therapy for ≥ 6 weeks, occurring within 6 months prior to Day 1 of study treatment.

Prior/Concomitant Therapy

* Patients receiving regularly scheduled blood (RBC) transfusion therapy (also termed chronic, prophylactic, or preventive transfusion)
* Receiving or use of concomitant medications that are strong inducers of CYP3A4/5 within 2 weeks of starting study treatment or anticipated need for such agents during the study
* Use of voxelotor within 28 days prior to starting study treatment or anticipated need for this agent during the study
* Use of an experimental selectin antagonist (eg, monoclonal antibody or small molecule) within 28 days of starting study treatment or anticipated need for such agents during the study
* Use of erythropoietin or other hematopoietic growth factor treatment within 28 days of starting study treatment or anticipated need for such agents during the study
* Receipt of prior cellular-based therapy (eg, hematopoietic cell transplant, gene modification therapy)

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2021-01-29 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2027-03-19 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin response rate | 24 Weeks
  Hemoglobin response rate at Week 24 (increase of > 1 g/dL [> 10 g/L] from baseline) during the blinded treatment period
Annualized vaso-occlusive crisis | 52 Weeks
  Annualized vaso-occlusive crisis rate during the 52-week blinded treatment period based on adjudicated vaso-occlusive crisis review

SECONDARY OUTCOMES:
Hemoglobin | 52 Weeks
  Change from baseline in hemoglobin at Week 52 during the blinded treatment period
Absolute reticulocyte count | 24 Weeks
  Change in absolute reticulocyte count from baseline at Week 24 during the blinded treatment period
Indirect bilirubin | 24 Weeks
  Change in unconjugated bilirubin from baseline at Week 24 during the blinded treatment period
Lactate dehydrogenase | 24 Weeks
  Change in lactate dehydrogenase from baseline at Week 24 during the blinded treatment period
Vaso-occlusive crisis | 52 Weeks
  Time to first vaso-occlusive crisis during the blinded treatment period
Fatigue | 52 Weeks
  Change in Patient-Reported Outcome Measurement Information System (PROMIS) Fatigue Scale from baseline in adult patients at Week 52 during the blinded treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (141):
- United States (63):
  - Univ of Alabama Birmingham, Birmingham, Alabama
  - Phoenix Children's Hsptl, Phoenix, Arizona
  - [Legal] Woodland International Research Group, LLC, Little Rock, Arkansas
  - [Legal] Collaborative Neuroscience Network, LLC, Long Beach, California
  - Pacific Research Partners, Oakland, California
  - UCSF Oakland Benioff ChildHosp, Oakland, California
  - University Of California Irvine, Orange, California
  - UC Davis Medical Center, Sacramento, California
  - University of Connecticut, Farmington, Connecticut
  - Yale University, New Haven, Connecticut
  - Howard University, Washington D.C., District of Columbia
  - Cornerstone Research Institute, Altamonte Springs, Florida
  - University of Florida, Gainesville, Florida
  - Foundation for Sickle Cell Disease Research, Hollywood, Florida
  - University Of Miami, Miami, Florida
  - Advanced Pharma CR, Miami, Florida
  - Arnold Palmer Children's Hospital, Orlando, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Sonar Clinical Research, Atlanta, Georgia
  - Children's Healthcare of Atlanta Investigational Medication Pharmacy, Atlanta, Georgia
  - Center for Blood Disorders Augusta University, Augusta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Children's Hosp-New Orleans, New Orleans, Louisiana
  - University Of Maryland School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital_Boston, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - [Legal] Dr. Vince Clinical Research, LLC and Dr. Vince Clinical Research, P.A., Detroit, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine_St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Children's National Health Hospital, Washington, New Jersey
  - NYC Health+Hospitals, Brooklyn, New York
  - Queens Hospital Center, Jamaica, New York
  - North Shore Long Island Jewish Medical Center, New Hyde Park, New York
  - Columbia University Medical Center_New York, New York, New York
  - Weill Cornell Med Coll-NYPH, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - [Legal] The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - [Legal] Children's Hospital Medical Center dba Cincinnati Children's, Cincinnati, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Neuro-Behavioral Clinical Research, North Canton, Ohio
  - Jimmy Everest Cancer Hematology & Oncology, Oklahoma City, Oklahoma
  - Lynn Institute of Tulsa, Tulsa, Oklahoma
  - Children's Hosptl Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health-Upstate, Greenville, South Carolina
  - Methodist University Hospital, Memphis, Tennessee
  - [Legal] St. Jude Children's Research Hospital, Memphis, Tennessee
  - [Legal] Baylor College of Medicine, Houston, Texas
  - UT Health University of Texas, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Mary Bridge Children's Health, Tacoma, Washington
  - Versiti Blood Center of Wisconsin, Milwaukee, Wisconsin
- Canada (4):
  - Providence Hematolgy, Vancouver, British Columbia
  - The Hospital for Sick Children, Toronto, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - CHU Sainte-Justine Mother and Child University Hospital, Montreal, Quebec
- Egypt (5):
  - [Legal] Alexandria Clinical Research LLC, Alexandria
  - Cairo University, Cairo
  - Ain Shams University Hospital, Cairo
  - Al Kasr AL Aini Hospital, Cairo
  - Sydnawy University Hospital, Zagazig
- France (6):
  - Ap-Hp-Hopital Henri Mondor, Créteil
  - Hospices Civils de Lyon-Hopital Edouard Herriot, Lyon
  - Centre Hospitalier Universitaire de Montpellier-Hopital Saint-Eloi, Montpellier
  - GHR Mulhouse Sud-Alsace, Mulhouse
  - Ap-Hp-Hopital Robert Debre, Paris
  - Saint-Denis Hospital Center, Saint-Denis
- Germany (6):
  - Charité - Campus Virchow-Klinikum - Klinik für Pädiatrie mit Schwerpunkt Onkologie und Hämatologie, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsklinikum Freiburg-Zentrum für Kinder- und Jugendmedizin, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf - University Medical Center Hamburg-Eppendorf, Hamburg
  - Uniklinik Heidelberg - Klinik für Pädiatrische Onkologie, Hämatologie, Immunologie und Pneumologie, Heidelberg
  - Universitätsklinikum Regensburg, Regensburg
- Ghana (2):
  - Ghana Institute of Clinical Genetics, Korle Bu Teaching Hospital (KBTH), Accra
  - Kintampo Health Research Centre (KHRC), Kintampo, Ghana, Kintampo
- Greece (4):
  - General University Hospital of Patras, Pátrai, Larissa
  - Gen Hosp Athens Ippokrateio,B' Uni Clinic Internal Medicine, Athens
  - General Hospital Of Larissa Koutlibaneio And Triantafylleio - Thalassemia and SCD Unit, Larissa
  - 'Ippokrateio' General Hospital of Thessaloniki, Thessaloniki
- India (5):
  - K.J Somaiya Hospital and Research Centre, Mumbai, Maharashtra
  - Yashoda Hospital, Hyderabad, Telangana
  - Victoria Hospital, Bangalore, Bangalore
  - Srirama Chandra Bhanj Medical College & Hospital (S.C.B Medical College), Cutack
  - All India Institute of Medical Sciences (AIIMS), New Delhi
- Italy (6):
  - Centro per lo Studio e la Cura delle Amiloidosi Sistemiche Fondazione IRCCS Policlinico San Matteo, Pavia, PV
  - Azienda Ospedaliero Universitaria Policlinico G. Rodolico - San Marco, Catania
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga - S.C.D.O. Microcitemie e malattie rare ematologiche, Orbassano
  - Azienda Ospedale Universita Padova, Padua
  - ARNAS Ospedali Civico Di Cristina Benfratelli - Presidio Ospedaliero "Civio e Benfratelli", Palermo
  - Ospedale Pediatrico Bambino Ges, Roma
- Kenya (4):
  - Kombewa Clinical Research Centre, Kisumu
  - KEMRI Kondele Children Hospital, Kisumu, Kisumu
  - KEMRI Siaya Clinical Research Annex Siaya County Referral Hospital, Siaya, Kisumu
  - Gertrude's Children's Hospital, Nairobi, Nairobi
- Lebanon (3):
  - Master Centre for Lebanon, Amman
  - American University of Beirut Medical center, Beirut
  - Hospital Nini, Tripoli
- Nigeria (5):
  - University of Abuja Teaching Hospital, Gwagwalada, Abuja, Abuja
  - Barau Dikko Teaching Hospital, Kaduna, Kaduna
  - Aminu Kano Teaching Hospital (AKTH), Kano
  - Lagos University Teaching Hospital, Lagos, Lagos
  - University of Nigeria Teaching Hospital, Enugu, Lagos
- Sultan Qaboos University Hospital, Muscat, Sultanet of Oman/Muscat/Al Khoud, Oman
- Saudi Arabia (3):
  - King Fahad Specialist Hospital-Dammam, Dammam
  - Prince Mohammad Bin Naser Hospital, Jizan
  - King Khaled University Hospital,King Saud Univ. Med. City, Riyadh
- Spain (10):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
- Turkey (Türkiye) (7):
  - Çukurova Üniversitesi Tıp Fakültesi Balcalı Hastanesi- Hematoloji, Adana
  - Başkent Üniversitesi Adana Dr. Turgut Noyan Uygulama ve Araştırma Merkezi, Adana
  - Adana City Training and Research Hospital, Adana
  - Hacettepe Üniversitesi Hastanesi- Hematoloji, Ankara
  - Ege Üniversitesi Tip Fakultesi Hastanesi - Nefroloji, Izmir
  - Mersin Üniversitesi Tip Fakültesi Hastanesi- Çiftlikköy Yerleşkesi- Hematoloji, Mersin
  - VM Medical Park Mersin Hastanesi- Kardiyoloji, Mersin
- United Kingdom (7):
  - Leicester Royal Infirmary - Haemostasis & Thrombosis Unit, Leicester
  - University Hospital Lewisham, Lewisham and Greenwich NHS Trust, London
  - Guys and St Thomas NHS Foundation Trust / Evelina Childrens Hospital, London
  - Kings College Hospital - Haematology, London
  - Hammersmith Hospital - London, London
  - Churchill Hospital, Oxford
  - Royal Hallamshire Hospital, Sheffield

REFERENCES:
- [Derived] Obadina M, Wilson S, Derebail VK, Little J. Emerging Therapies and Advances in Sickle Cell Disease with a Focus on Renal Manifestations. Kidney360. 2023 Jul 1;4(7):997-1005. doi: 10.34067/KID.0000000000000162. Epub 2023 May 31. PMID 37254256
- [Derived] Forsyth S, Schroeder P, Geib J, Vrishabhendra L, Konstantinidis DG, LaSalvia K, Ribadeneira MD, Wu E, Kelly P, Kalfa TA. Safety, Pharmacokinetics, and Pharmacodynamics of Etavopivat (FT-4202), an Allosteric Activator of Pyruvate Kinase-R, in Healthy Adults: A Randomized, Placebo-Controlled, Double-Blind, First-in-Human Phase 1 Trial. Clin Pharmacol Drug Dev. 2022 May;11(5):654-665. doi: 10.1002/cpdd.1058. Epub 2022 Jan 12. PMID 35019238